CLINICAL TRIAL: NCT00725972
Title: Pre-emptive Hemodynamic Optimization of High Risk Patients Undergoing Elective Major Surgical Procedures.
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: termination of funding by sponsors
Sponsor: University of Pittsburgh (Other)
Collaborators: Hutchinson Technology Inc (Industry); Cheetah Medical Inc. (Industry); LIDCO Limited (Unknown)
Responsible Party: Principal Investigator, Hernando Gomez, Assistant Professor, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: Goal Directed Therapy
Record Dates: First submitted 2008-07-22; First posted 2008-07-31 (Estimated); Last update posted 2017-08-01 (Actual); Status verified 2017-07

CONDITIONS: Hemorrhage
Keywords: Improve; Patient care; Applying; Systematic; Fashion; Proven; Resuscitation; Algorithms; High risk; Surgical
MeSH Terms: conditions — Hemorrhage

STUDY DESIGN:
Intervention Model Description: A protocol group receiving augmented Oxygen Delivery will be compared to a usual care group.
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants undergo anesthesia and are unaware of the arm they are in. Outcomes Assessors are only given data on results and are kept unaware of the peri-operative management.
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Augmented Oxygen Delivery Group (Experimental): Hemodynamic management to a goal of O2 delivery of 600 ml/m2/min utilizing cardiac stroke volume variation with positive pressure ventilation to optimize fluid management.
  Intervention: Augment O2 Delivery by hemodynamic protocol. (7/30/17: deleted original text which apparently was pasted from an entirely unrelated study having to do with age of transfused blood, presumably by the creator of this record, Cynthia Hatfield, in 2010. SLW)
  Interventions: Other: Augment O2 Delivery by hemodynamic protocol
- Control (Sham Comparator): Patients having the same types of surgery but receiving usual anesthetic care. Intervention: High Risk Surgery. (7/30/17: deleted original text which apparently was pasted from an entirely unrelated study having to do with age of transfused blood, presumably by the creator of this record, Cynthia Hatfield, in 2010. SLW)
  Interventions: Procedure: High Risk Surgery

INTERVENTIONS:
Other: Augment O2 Delivery by hemodynamic protocol — Hemodynamic management to a goal of O2 delivery of 600 ml/m2/min utilizing cardiac stroke volume variation with positive pressure ventilation to optimize fluid management.
  Arms: Augmented Oxygen Delivery Group
Procedure: High Risk Surgery — Patients with same characteristics as Experimental Group having same types of Surgery but no change to usual anesthetic care
  Arms: Control

SUMMARY:
Several recent clinical trials have documented that early aggressive resuscitation approached guided by defined hemodynamic variables using thoughtful protocols may improve outcome. The concept underscored by this newer trial was that appropriate resuscitation prevents subsequent tissue injury even if overt shock is present, if the resuscitation is carried out early enough.

DETAILED DESCRIPTION:
This is a randomized, prospective study which will include a total of 200 patients who are scheduled to undergo major elective surgery with an anticipated blood loss of ≥ 500 ml. The research participants will be randomly assigned to a control group (n=100) that will receive the standard of care for intraoperative management by the anesthesia. Minimal resuscitation standards include a mean arterial pressure > 65 mm Hg, SpO2 > 90% and evidence of end-organ perfusion (i.e. mentation prior to induction of anesthesia, urine output > 20 ml/hr) and absence of tachycardia (HR < 100/min). The protocol group (n=100) will, in addition, receive further resuscitation to achieve an increased oxygen delivery (DO2) to a targeted of 600 ml/min/m2. This approach is called goal-directed therapy. This target DO2 will be achieved via a treatment algorithm that includes intraoperative volume expansion and/or dobutamine infusion, guided by the LiDCO cardiovascular monitoring of stroke volume and cardiac output. All patients will also have non-invasive tissue O2 saturation (StO2) monitoring using the InSpectra probe on their hand. Patients in the protocol group will be subdivided to 2 subgroups. Group one subjects will be those patients that are directly admitted to the ICU following surgery and group two subjects will be those patients discharged to the PAR and then a regular hospital ward. All subjects will continue to receive goal directed therapy for as long as they are in the PAR or ICU or until 8 hours of post-operative time has elapsed. All participants will be followed daily during their hospital stay to assess the development of complications, length of stay and discharge status. All patients will receive phone interview at one and 3 months after the surgery to inquire about their quality of life since their surgery using the SF36 instrument. The total duration of participant's commitment to the study will be 3 months, during which their lab and clinical data will be recorded. Statistical analysis of the data will be performed at the conclusion of the study period by professional statistician to determine the difference in the outcome and morbidity and mortality between the two groups using multiple logistic regression and Cox proportional hazard scoring with primary outcome variables being length of stay, total complications, and mortality.

ELIGIBILITY:
Inclusion Criteria:

* Adult, Male or female.
* Patients undergoing elective major surgery.
* Patients with normal renal function.
* All patients will sign informed consent.

Exclusion Criteria:

* Major organ failure.
* Low cardiac output conditions.
* Pulmonary hypertension.
* Severe pulmonary disease.
* Patient refusal to participate in the study.
* Pregnancy.
* Emergency Surgery.
* Lithium allergy or patient on lithium.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2008-07 (Actual)

PRIMARY OUTCOMES:
Duration of mechanical ventilation. Duration of ICU and hospital stay. Infection Renal function. Bowel movement. Oral intake. 3-month period Quality of life. | 3 months

SECONDARY OUTCOMES:
As in the primary | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Steven L Whitehurst, MD, Principal Investigator — University of Pittsburgh Medical Center
Locations (1):
- UPMC-Presbyterian Hospital, Pittsburgh, Pennsylvania, United States